CLINICAL TRIAL: NCT06778993
Title: Using a Wearable Breast Simulator Breastfeeding Education Provided to Pregnant Women and Their Wives Mothers' Perceived Partner Support, Breastfeeding Self-Efficacy and Determining the Influence of Fathers on Breastfeeding
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rasime Yıldırım Dugeroglu, Lecturer, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Date 04.04.2023/decision no.07
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Breastfeeding
Keywords: breastfeeding; wearable breast simulator; nursing; father; mother; Breastfeeding Self-Efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The implementation will begin in the clinic, where the researcher will administer an introductory form to couples in their 34th-36th weeks of pregnancy. Depending on the group assignments, participants will either receive breastfeeding education with a simulator or proceed without intervention. The process will continue in the hospital during the 38th-40th weeks of pregnancy, followed by postpartum visits on days 1-3 at participants' homes. Further monitoring will be conducted during the 1st and 6th weeks postpartum at their homes. The monitoring form and the designated scales will be completed face-to-face by the researcher during these visits.
  Interventions: Other: Breastfeeding Education Program Accompanied by a Wearable (Hybrid) Simulator
- Controlled Group (No Intervention): There is no intervention.

INTERVENTIONS:
Other: Breastfeeding Education Program Accompanied by a Wearable (Hybrid) Simulator — This training is conducted in both theoretical and practical formats. The theoretical training consists of two sessions, each lasting 25 minutes, with a 10-minute break in between, totaling 60 minutes. Following the theoretical training, simulation-based skill training is conducted. This phase also comprises two sessions of 25 minutes each, with a 10-minute break, making a total duration of 60 minutes.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate the impact of breastfeeding education using a wearable breast simulator on perceived spousal support, breastfeeding self-efficacy, and breastfeeding outcomes in pregnant women and their spouses. The main questions it aims to answer are:

Does education with a wearable breast simulator improve mothers' breastfeeding self-efficacy and perceived spousal support compared to standard education? Does this intervention positively influence fathers' involvement in breastfeeding and overall breastfeeding outcomes? Researchers will compare participants receiving the wearable simulator-based breastfeeding education to those receiving standard care to determine its effects on these outcomes.

Participants will:

Complete demographic and pre-test questionnaires, including breastfeeding self-efficacy and spousal support scales.

Attend two 25-minute theoretical and two 25-minute simulation-based training sessions using a wearable breast simulator.

Fathers will practice breastfeeding techniques, including baby positioning and milk expression, with the simulator.

Postpartum, participants will be assessed at the hospital and during follow-ups at home (1st and 6th weeks) for changes in perceived spousal support, breastfeeding self-efficacy, and fathers' involvement in breastfeeding.

DETAILED DESCRIPTION:
Breastfeeding Education Given to Pregnant Women and Their Partners Using a Wearable Breast Simulator on Mothers' Perceived Spousal Support, Breastfeeding Self-Efficacy and Fathers' Breastfeeding. In this training, it is planned to provide training and implementation to pregnant women and their partners who have no previous breastfeeding experience .

The training is given theoretically to mothers and fathers, and the fathers-to-be are also given some practical experience and are made to wear a simulator.

In the study, women;

* Their perceived spousal support is high,
* Only the mother networks have a long data delivery time,
* Having a high level of breastfeeding self-efficacy,
* The aim is to have a positive effect on fathers' breastfeeding. Purpose of the research The aim of this study is to evaluate the effects of breastfeeding education provided during the prenatal period by wearing the breast on mother and father days, on perceived spousal support, the effect of breastfeeding on fathers' breastfeeding, and the reproductive effects of breastfeeding in the postnatal period.

Data Collection: The implementation will commence in the clinic by the researcher with the administration of an introductory form to couples in their 34th-36th weeks of pregnancy. Subsequently, based on the groups, participants will either receive breastfeeding education using a simulator or proceed without intervention. The process will continue during the 38th-40th weeks of pregnancy at the hospital, followed by postpartum home visits on days 1-3, and in the 1st and 6th weeks. During these visits, the monitoring form and the designated scales will be administered face-to-face by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* The expectant mother has a contraindicated condition for breastfeeding, The mother has a mental disability or a severe psychiatric disorder, The expectant mother has not received planned, professional breastfeeding education with her partner during pregnancy, The mother has communication issues.

Exclusion Criteria:

* The newborn has a health issue that prevents breastfeeding, During the follow-up process of the study, the couple cannot be reached for any reason using the communication information provided, Premature birth (before the 37th week of pregnancy), A situation arises post-birth that prevents the mother, father, and baby from being together, The newborn has a health condition that hinders or negatively affects breastfeeding, The death of the mother and/or father, The development of a health issue in the mother that could prevent breastfeeding (such as breast cancer, severe heart disease), Participants choosing to withdraw from the study voluntarily.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-03-24 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 34th-36th Weeks of Pregnancy, 38th-40th Weeks of Pregnancy, Postpartum Days 1-3, 1st Week, and 6th Week
  To determine the characteristics to be utilized in the study, the researcher prepared two separate introductory forms for mothers and fathers by reviewing the relevant literature.
  The mother's introductory form includes sections on the sociodemographic characteristics of the expectant mother, information related to pregnancy, breastfeeding, and breast milk, as well as postpartum-specific details, including sections on the mother's characteristics during the 1st to 6th weeks postpartum.
  The father's introductory form covers the sociodemographic characteristics of the expectant father, his knowledge and perspectives regarding pregnancy and the breastfeeding process, the father's relationship with the mother and baby during the postpartum period, and the father-baby relationship during the 1st to 6th weeks postpartum.
Short Form of the Antepartum-Postpartum Breastfeeding Self-Efficacy Scale | 34th-36th Weeks of Pregnancy, 38th-40th Weeks of Pregnancy, Postpartum Days 1-3, 1st Week, and 6th Week
  The Breastfeeding Self-Efficacy Scale was developed by Dennis in 1999 and consists of 33 items. Initially, it was applied to 130 English-speaking Canadian women, yielding a Cronbach's alpha value of 0.96, with 73% of the items having item-total correlations ranging from 0.30 to 0.70. In 2003, Dennis revised the scale, reducing it to a 14-item version, creating the Short Form of the Breastfeeding Self-Efficacy Scale. The short form is a 5-point Likert scale, with responses ranging from 1 ("Not sure at all") to 5 ("Always sure"). AThe minimum score obtainable is 14, and the maximum score is 70. A higher score indicates higher breastfeeding self-efficacy.
Father's Impact on Breastfeeding Scale | 34th-36th Weeks of Pregnancy, 38th-40th Weeks of Pregnancy, Postpartum Days 1-3, 1st Week, and 6th Week
  The Father's Impact on Breastfeeding Scale, consisting of 37 items, evaluates how frequently fathers engage in activities while the mother is breastfeeding, using a Likert-type rating scale from 1 to 5. Each item is scored on a 5-point Likert scale, where 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, and 5 = Very Often. The scale contains five subdimensions: understanding breastfeeding, assistance, appreciation, availability, and sensitivity.A higher total score on the scale indicates a greater impact of fathers on breastfeeding. The minimum score that can be obtained from the scale is 37, while the maximum score is 185.
Perceived Partner Support Scale in the Early Postpartum Period | 34th-36th Weeks of Pregnancy, 38th-40th Weeks of Pregnancy, Postpartum Days 1-3, 1st Week, and 6th Week
  The Perceived Partner Support Scale in the Early Postpartum Period, developed in a 5-point Likert format, aims to determine the level of perceived partner support during the early postpartum period. The scale contains both positive and negative statements mixed together. The positive items are 1, 2, 3, 4, 5, 6, 7, 11, 13, and 16, while the negative items are 8, 9, 10, 12, 14, and 15.The highest possible score on the scale is 80, and the lowest possible score is 16.

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Şenturk Erenel, Study Director — Lokman Hekim University
Locations (1):
- Private Obstetrics Clinics in Kırşehir Province, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No